CLINICAL TRIAL: NCT00295165
Title: Randomized, Double-Blind, Placebo-Controlled, Phase 3 Induction Study to Assess the Efficacy and Safety of 6µg Sargramostim (Leukine) Administered Subcutaneously Once Daily for 8 Weeks in Patients With Active Crohn's Disease
Brief Title: Efficacy (Induction of Response/Remission) and Safety Study in Patients With Moderate to Severe Crohn's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 310187; 91494; NOVEL8; NCT00295321 (obsolete NCT alias)
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — sargramostim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Sargramostim (Leukine)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sargramostim (Leukine) — Sargramostim 6 mcg/kg subcutaneously once daily
  Other Names: BAY86-5326
  Arms: Arm 1
Drug: Placebo — Placebo subcutaneously once daily
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate if Leukine can induce clinical response or remission in patients with Crohn's disease.

DETAILED DESCRIPTION:
On 29 May 2009, Bayer began transitioning the sponsorship of this trial to Genzyme. NOTE: This study was originally posted by sponsor Berlex, Inc. Berlex, Inc. was renamed to Bayer HealthCare, Inc.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Male or female, age >/= 18 years
3. Confirmed diagnosis of Crohn's disease (endoscopic or radiological evaluation) at least 4 months prior to receiving the first dose of study drug
4. Moderately to severely active Crohn's disease at time of screening (i.e., CDAI greater than or equal to 220 and less than or equal to 475 points)
5. If under treatment for Crohn's disease, medication must be stable for at least 4 weeks prior to receiving the first dose of study drug. The following therapies are allowed:

   * Oral therapy with salicylates (mesalamine, sulfasalazine, olsalazine, or balsalazide) for Crohn's disease
   * Antibiotics or probiotics for Crohn's disease
   * Topical rectal therapy with mesalamine
6. Females of child-bearing potential:

   Negative pregnancy test within 72 hours prior to receiving the first dose of study drug
7. Sexually-active males and females of child-bearing potential:

   Agreement to use adequate method of contraception throughout the study
8. Ability to self-inject study drug or availability of a designee who can do so

Exclusion Criteria:

1. Pregnancy or breast-feeding
2. Colostomy or ileostomy
3. Immediate need for gastrointestinal (GI) surgery for active GI bleeding, peritonitis, intestinal obstruction, or intra-abdominal or perianal abscess requiring surgical drainage
4. GI surgery within 6 months prior to receiving the first dose of study drug
5. Symptoms of bowel obstruction or confirmed evidence of a clinically-significant stricture within the last 6 months that has not been surgically corrected
6. Positive stool test results for any of the following:

   Bacteria:
   * Salmonella spec.
   * Shigella spec.
   * Campylobacter spec.

   Bacterial toxin:
   * Clostridium difficile

   Ova and parasites:
   * Amoeba spec.
   * Giardia spec.
   * Cryptosporidium spec.
7. Any of the following laboratory abnormalities:

   * Serum creatinine >/= 2.0 mg/dL
   * Alkaline phosphatase (AP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin >/=; 2 x the upper limit of normal
   * Hemoglobin (Hgb) < 8.0 g/dL
   * Absolute neutrophil count (ANC) </= 1,000 cells/µL or > cells 20,000/µL
8. Planned in-patient hospitalization during the study
9. Presence or history of cancer of any type (except treated basal cell carcinoma) or definite dysplasia of the colon within the last 5 years
10. Use of any of the following medications during the specified period of time prior to receiving the first dose of study drug:

    At any time:
    * Recombinant human GM CSF (sargramostim or molgramostim)
    * Granulocyte colony-stimulating factor (G CSF; filgrastim or pegfilgrastim)
    * Natalizumab 8 weeks: or 5 half-lives (whichever is longer)
    * Licensed/registered and/or experimental anti-tumor necrosis factor (TNF) therapy such as infliximab or adalimumab 4 weeks:
    * 6-mercaptopurine
    * Azathioprine
    * Cyclophosphamide
    * Methotrexate
    * Mycophenolate mofetil
    * Tacrolimus
    * Cyclosporine
    * Thalidomide
    * Glucocorticoids, including budesonide and prednisone, or local glucocorticoid therapy for Crohn's disease
    * Any other immunosuppressive drugs
11. Use of any investigational drug within 4 weeks or 5 half-lives (whichever is longer) prior to receiving the first dose of study drug
12. Use of nutritional therapy (parenteral nutrition or enteral nutrition with elemental or semi-elemental diets) within 4 weeks prior to receiving the first dose of study drug. If the physician judges that nutritional supplementation is needed, enteral nutritional supplements will be allowed for patients who have been receiving a stable regimen for at least 4 weeks prior to receiving the first dose of study drug and that is intended to continue through the 8 week treatment period.
13. History of allergy to yeast products or to sargramostim or to any other excipient of the study drug formulation
14. Active drug or alcohol abuse
15. Clinically important co-morbid conditions unrelated to Crohn's disease as determined by the investigator
16. Previous randomization into this study, or into any other study of the sponsor's sargramostim development program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-01; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To induce clinical remission and/or clinical response following 8 weeks of treatment | 8 weeks

SECONDARY OUTCOMES:
To assess the safety profile of sargramostim (including development of antibodies against sargramostim) | During study treatment
To assess quality of life (QoL) | During study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (98):
- United States (46):
  - Huntsville, Alabama
  - Orange, California
  - San Francisco, California
  - Lakewood, Colorado
  - Littleton, Colorado
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Gainesville, Florida
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Hagerstown, Maryland
  - Lutherville, Maryland
  - Towson, Maryland
  - Ann Arbor, Michigan
  - Chesterfield, Michigan
  - Troy, Michigan
  - Plymouth, Minnesota
  - Mexico, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Florham Park, New Jersey
  - New Brunswick, New Jersey
  - Great Neck, New York
  - Mineola, New York
  - New York, New York
  - Syracuse, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Sayre, Pennsylvania
  - Columbia, South Carolina
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Chesapeake, Virginia
  - Christiansburg, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Wenatchee, Washington
- Australia (8):
  - Liverpool, New South Wales
  - Caboolture, Queensland
  - Adelaide, South Australia
  - Frankston, Victoria
  - Melbourne, Victoria
  - Brisbane
  - Hamilton
  - Sydney
- Brazil (5):
  - Blumenau, Santa Catarina
  - Florianópolis, Santa Catarina
  - Botucatu, São Paulo
  - São Paulo, São Paulo
  - Santos
- Bulgaria (2):
  - Sofia
  - Varna
- Canada (10):
  - Abbotsford, British Columbia
  - Winnipeg, Manitoba
  - Saint John, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Guelph, Ontario
  - Kingston, Ontario
  - Ottawa, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Saint-Charles-Borromée, Quebec
- Israel (5):
  - Haifa, Israel
  - Ẕerifin, Israel
  - Jerusalem
  - Rehovot
  - Tel Aviv
- New Zealand (4):
  - Auckland
  - Dunedin
  - Hamilton
  - Tauranga
- Romania (2):
  - Bucharest
  - Craiova
- Russia (4):
  - Kazan'
  - Krasnodar
  - Moskva
  - Saint Petersburg
- South Africa (6):
  - Port Elizabeth, Eastern Cape
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Cape Town, Western Cape
  - Somerset West, Western Cape
  - Durban
- Ukraine (6):
  - Dnipro
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Lviv
  - Zaporizhzhya